CLINICAL TRIAL: NCT04394728
Title: Research of Serum and Urine Metabolomic Biomarkers Predictive Pharmacokinetic Parameters of Trabectidin in Patients With Soft Tissues Sarcomas
Brief Title: Pharmacometabolomic of Trabectedin in Soft Tissue Patients
Acronym: Metabol-STS
Status: Completed | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2015-04
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Sarcoma
Keywords: soft tissues sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Trabectedin — 1.3 mg/m2 with a top-dose of 2.6 mg per cycle, via a central venous catheter as a 24-hour infusion every 21 days.All patients received premedication with dexamethasone 20 mg i.v. 30 min before administration of trabectedin.
  Other Names: Yondelis

SUMMARY:
This perspective, mono institutional study is addressed to find potential serum and urine biomarkers predictive of the pharmacokinetic and pharmacodynamic profile of soft tissue sarcomas patients treated with trabectedin.

DETAILED DESCRIPTION:
This investigation enrolled patients with unresectable and/or metastatic soft tissue sarcoma not responsive to the first-line treatment based on anthracycline/ifosfamide. Patients underwent trabectedin monotherapy that was administered intravenously at the dose of 1.3 mg/m2 every 21 days.

Single overnight fasting urine and blood samples were collected on day-1 of the first trabectedin administration.

Plasma pharmacokinetics was performed during cycle 1. Blood samples, drawn from a site separate from the drug infusion site, were obtained prior to the infusion (basal) at 2, 8, 24 (end of infusion) and 0.5, 1.0, 4.0, 8.0, 24.0 after the end of the infusion. Plasma concentrations of trabectedin were measured by liquid chromatography, tandem mass spectrometry assay (LC-MS/MS) and the pharmacokinetic parameters (Cmax, Clearance, AUC and T1/2) were calculated from the concentration-time curve using a non-compartmental model.

Metabolomics profiles were explored by LC-MS/MS in predose urine and serum and encompassed a total of 192: a) 45 amino acid derivatives, virtually involved in a wide set of biochemical pathways; b) 40 different acylcarnitines, principally involved in the cellular energy metabolism; c) 15 lysophosphatidylcholine metabolites, 77 phosphatidylcholine derivatives, and 15 sphingomyelins, involved in fatty acid metabolism and cellular signaling. The identification of predictive metabolomics biomarkers is performed using univariate and multivariate statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Soft Tissues Sarcoma STSs (unresectable and/or metastatic disease).
* One previous systemic treatment with ananthracycline ± ifosfamide.
* Measurable disease, as defined by RECIST criteria.
* ECOG PS ≤2.
* Age ≥18 years.
* A minimum of 3 weeks since prior tumor directed therapy
* Recovery from toxic effects of prior therapies to NCI CTC Grade 1 or lower.
* Adequate haematological, renal liver function.
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women
* Prior exposure to Trabectedin.
* Peripheral neuropathy, Grade 2 or higher.
* Known CNS metastases.
* Active viral hepatitis or chronic liver disease.
* Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within one year before enrolment, uncontrolled arterial hypertension or arrhythmias.
* Active major infection.
* Other serious concomitant illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Soft tissue sarcoma patients with unresectable and/or metastatic disease
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | 0-48 hours
  Pharmacokinetics profile of Trabectedin for 24 hours intravenous infusion
Cmax | 0-48 hours
  Maximum plasma concentration of Trabectedin
Metabolomics profile | 0 hours ( pre-dose)
  Predose metabolomic profile in serum and urine

SECONDARY OUTCOMES:
Progression free survival | 2 years
  From the first day of treatment to progression or death due to any cause
Overall survival | 2 years
  The time from the first course of trabectedin to death from any cause or to the last follow-up
Treatment Toxicity | through study completion, an average of 1 year
  Hematologic and non-hematologic toxicity according to WHO

CONTACTS AND LOCATIONS:
Overall Officials: Gianmaria Miolo, Principal Investigator — Centro di Riferimento Oncologico - Aviano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pharmaco-metabolomics: An Emerging "Omics" Tool for the Personalization of Anticancer Treatments and Identification of New Valuable Therapeutic Targets — https://pubmed.ncbi.nlm.nih.gov/22105661/